CLINICAL TRIAL: NCT02280863
Title: Hybrid Closed-Loop Studies With Medtronic PID Controller- Hotel HCL Study
Brief Title: Hybrid Closed-Loop Hotel Studies With Medtronic PID Controller
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Bruce A. Buckingham, Principle Investigator, Stanford University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IDE: G140086; 1-SRA-2014-238- (Other Grant/Funding Number: JDRF Grant Key: 1-SRA-2014-238-M-R); IRB 29973 (Other: Stanford University)
Record Dates: First submitted 2014-07-09; First posted 2014-11-03 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adult Cohort (Experimental): Medtronic Hybrid Closed-Loop System will be used by adults for five days in open-loop (sensor augmented pump) and five days in closed-loop. The first 8 Adults use the Android Platform.
  Interventions: Device: Medtronic Hybrid Closed-loop System - Android Platform; Device: Medtronic Hybrid Closed-loop Integrated System
- Adolescent Cohort (Experimental): Medtronic Hybrid Closed-Loop System will be used by adolescents for four days in open-loop (sensor augmented pump) and four days in closed-loop.
  Interventions: Device: Medtronic Hybrid Closed-loop Integrated System

INTERVENTIONS:
Device: Medtronic Hybrid Closed-loop System - Android Platform — A continuous glucose sensor and insulin delivery system designed for continuous closed-loop control with the PID-IFB (proportional-integral-derivative insulin feed-back) algorithm using an Android controller.
  Arms: Adult Cohort
Device: Medtronic Hybrid Closed-loop Integrated System — A fully integrated continuous glucose sensor and insulin delivery system designed for continuous closed-loop control with the PID-IFB (proportional-integral-derivative insulin feed-back) algorithm

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of the Medtronic hybrid closed-loop (HCL) system utilizing the proportional-integral-derivative algorithm with insulin feedback (PID-IFB) optimized to function in a hybrid mode with closed-loop control operating during the day and night.

DETAILED DESCRIPTION:
Study participants will be asked to use the CGM and the study insulin pump provided for approximately 4 to 5 days prior to initiation of the HCL PID-IFB system in a hotel setting for another 4 to 5 days. All participants with diabetes and the parent/ guardian of participants < 18 years of age will be asked to stay overnight in a hotel while the HCL PID-IFB system is on and to remain close to Stanford University during the day. For participants > 18 years of age, designated remote monitors will be asked to receive alerts for low/ high glucose levels.

Enrolled participants will be asked to complete evaluations to describe their user experience/ evaluation of the system.Each participant had a companion (parent/ legal guardian of participants < 18 years of age, or the designate remote monitor for participants > 18 years of age) who will consent to monitor the participant and complete an evaluation, but will not be considered enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes (The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.)
* Daily insulin therapy for at least one year
* Age between 14.0 to 40.0 years of age. The first 9 subjects (between all 3 centers) will be over 18 years old.
* Subject has performed an average of at least 3 meter glucose readings per day in the preceding 2 weeks
* Subject has used a downloadable insulin pump for at least 3 months
* Subject comprehends written English
* Female patients who are sexually active must be on acceptable method of contraception e.g. oral contraceptive pill, diaphragm, IUD
* Female patients must have a negative urine pregnancy test
* Informed Consent Form signed by the subject and/or parent and assent signed by the subject if < age 18
* Parent/guardian (for subjects < 18 years) and subject understand the study protocol and agree to comply with it. Both parents must sign if possible.
* Total daily insulin requirement greater than 0.4 units/kg/day over the preceding two weeks.
* No expectation that subject will be moving out of the area of the clinical center during the study.
* Adults will need to be working within 20 minutes of our research staff during the day.
* A person willing to fulfill the role of a remote monitor (such as parent, spouse or significant other).

Exclusion Criteria:

* Subject has a medical disorder that in the judgment of the investigator will affect the wearing of the devices or the completion of any aspect of the protocol
* Diabetic ketoacidosis in the past month
* History of seizure or loss of consciousness in the last 6 months
* Subject has a respiratory condition such as asthma, treated with systemic or inhaled corticosteroids in the previous 6 months or cystic fibrosis
* Subject has a history of any cardiac or vascular disorder such as myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, arrhythmia or thromboembolic disease
* Subject has a history of liver or kidney disease (other than microalbuminuria)
* Systolic blood pressure > 140 mmHg on screening visit
* Diastolic blood pressure > 90 mmHg on screening visit
* Subject has active Graves' disease
* Subjects with inadequately treated thyroid disease or celiac disease
* Subject has a neurologic disorder that in the judgment of the investigator will affect completion of the protocol
* Either the subject or the subject's primary caregiver has received inpatient psychiatric treatment in the past 6 months
* Subject has a history of diagnosed medical eating disorder
* Subject has a history of known illicit drug abuse
* Subject has a history of known prescription drug abuse
* Subject has a history of current alcohol abuse
* Subject has a history of visual impairment which would not allow subject to participate
* Subject has an active skin condition that would affect sensor placement
* Subject has adhesive allergies
* Subjects requiring an intermediate or long-acting insulin (such as NPH, detemir or glargine)
* Subjects requiring other anti-diabetic medications other than insulin (oral or injectable)
* Current use of oral/inhaled glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study
* Subject is currently on beta blocker medication
* Subject is currently participating in another investigational study (drug or device)
* Subject is deemed by the investigator to be unwilling or unable to follow the protocol

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Buckingham, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Stanford University Medical Center, Stanford, California
  - UC Denver- Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Yale University- Department of Pediatric Endocrinology, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
There were three sites involved with the study; de-identified information was shared with the Denver and Yale sites.

REFERENCES:
- [Result] Ly TT, Weinzimer SA, Maahs DM, Sherr JL, Roy A, Grosman B, Cantwell M, Kurtz N, Carria L, Messer L, von Eyben R, Buckingham BA. Automated hybrid closed-loop control with a proportional-integral-derivative based system in adolescents and adults with type 1 diabetes: individualizing settings for optimal performance. Pediatr Diabetes. 2017 Aug;18(5):348-355. doi: 10.1111/pedi.12399. Epub 2016 May 18. PMID 27191182
- [Derived] Adams RN, Tanenbaum ML, Hanes SJ, Ambrosino JM, Ly TT, Maahs DM, Naranjo D, Walders-Abramson N, Weinzimer SA, Buckingham BA, Hood KK. Psychosocial and Human Factors During a Trial of a Hybrid Closed Loop System for Type 1 Diabetes Management. Diabetes Technol Ther. 2018 Oct;20(10):648-653. doi: 10.1089/dia.2018.0174. Epub 2018 Sep 21. PMID 30239219

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults were recruited in the first 2 cohorts. Following analysis of the adult cohorts, adolescents were recruited in the third cohort.
Groups:
- Adult Cohort: In part 1, participants used the system with Android interface running the algorithm; in part 2, participants used the integrated system which ran the algorithm on the pump.
  Medtronic Hybrid Closed-Loop System used by adults for five days in open-loop (algorithm off; sensor augmented pump) and five days in closed-loop (algorithm on). Algorithm was the PID-IFB (proportional-integral-derivative insulin feed-back) algorithm.
- Adolescent Cohort: Participants only participated in part 2, which used the integrated system which ran the algorithm on the pump.
  Medtronic Hybrid Closed-Loop System used by adolescents for four days in open-loop (algorithm off; sensor augmented pump) and four days in closed-loop (algorithm on). Algorithm was the PID-IFB (proportional-integral-derivative insulin feed-back) algorithm.
Period: Android Platform
Arm/Group | Adult Cohort | Adolescent Cohort
Started | 8 | 0
Completed | 8 | 0
Not Completed | 0 | 0
Period: Integrated Platform
Arm/Group | Adult Cohort | Adolescent Cohort
Started | 9 (One additional participant was enrolled for part 2.) | 15
Completed | 9 | 14
Not Completed | 0 | 1
Not completed — Met stopping criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adult Cohort | Adolescent Cohort | Total
Number analyzed (Participants) | 9 | 15 | 24
Age, Customized [Count of Participants; unit: Participants]
  0-12 year | 0 | 0 | 0
  13-17 years | 0 | 15 | 15
  18-64 years | 9 | 0 | 9
  65 year and older | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 1 | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With no More Than One Meter Glucose Value <50 mg/dL and no Values <40 mg/dL, no More Than Two Episodes With Meter Glucose Values Remaining >300 mg/dL for More Than 1 Hour, and no Ketonemia, Seizures, or Loss of Consciousness
Description: Our definition of a subject successfully participating in a cohort is:
  1. No more than one meter glucose value <50 mg/dL and no values <40 mg/dL
  2. No more than two episodes with meter glucose values remaining >300 mg/dL for more than 1 hour that are unrelated to an infusion set failure
  3. No ketonemia >1.0 mmol/L, while the system is functional unless related to an intercurrent illness or infusion set failure
  4. No seizures or loss of consciousness while system is on and functional
Time Frame: Up to 10 days
Measure: Count of Participants; unit: Participants
Groups:
- Adult Cohort - Medtronic Android Interface; Adult Cohort - Integrated System Interface: In part 1, participants used the system with Android interface running the algorithm; in part 2, participants used the integrated system which ran the algorithm on the pump.
  Medtronic Hybrid Closed-Loop System used by adults for five days in open-loop (algorithm off; sensor augmented pump) and five days in closed-loop (algorithm on). Algorithm was the PID-IFB (proportional-integral-derivative insulin feed-back) algorithm.
Arm/Group | Adult Cohort - Medtronic Android Interface | Adult Cohort - Integrated System Interface | Adolescent Cohort
Number analyzed (Participants) | 8 | 9 | 15
Participants | 0 | 0 | 1

2. Secondary Outcome: Mean Glucose Values
Description: Mean glucose values are reported as assessed by continuous glucose monitoring (CGM; subcutaneous sensor, day and night values).
Time Frame: Up to 10 days
Population: Participants who completed the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Adult Cohort - Medtronic Android Interface | Adult Cohort - Integrated System Interface | Adolescent Cohort
Number analyzed (Participants) | 8 | 9 | 14
mg/dL
  Day (open loop) | 151 (14) | 144 (15) | 171 (30)
  Day (closed loop) | 156 (14) | 152 (14) | 153 (17)
  Night (open loop) | 156 (26) | 142 (18) | 168 (39)
  Night (closed loop) | 155 (22) | 148 (20) | 144 (19)

3. Secondary Outcome: Mean Glucose Values, Fingerstick Glucose Meter Value, Adult Cohorts
Description: Mean glucose values are reported as assessed by fingerstick glucose meter value.
Time Frame: Up to 10 days
Population: Data are presented for adult cohorts only.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Adult Cohort - Medtronic Android Interface | Adult Cohort - Integrated System Interface
Number analyzed (Participants) | 8 | 9
mg/dL
  Open loop | 148 (31) | 164 (41)
  Closed loop | 127 (14) | 151 (36)

4. Secondary Outcome: Median Glucose Values, Fingerstick Glucose Meter Value, Adolescent Cohort
Description: Median an glucose values are reported as assessed by fingerstick glucose meter value.
Time Frame: Up to 10 days
Population: Data are presented for the adolescent cohort only. Participants who completed the protocol were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Adolescent Cohort
Number analyzed (Participants) | 14
mg/dL
  Open loop | 181 [121 to 191]
  Closed loop | 132 [121 to 138]

5. Secondary Outcome: Percentage of Time Within Glucose Range of 70-180 mg/dL
Time Frame: Up to 10 days
Population: Participants who completed the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of time in range
Arm/Group | Adult Cohort - Medtronic Android Interface | Adult Cohort - Integrated System Interface | Adolescent Cohort
Number analyzed (Participants) | 8 | 9 | 14
percentage of time in range
  Open loop | 71.9 (10.6) | 67.7 (8.1) | 55.2 (14.2)
  Closed loop | 71.0 (12.4) | 71.8 (12.5) | 69.8 (9.7)

6. Secondary Outcome: Percentage of Fingerstick Meter Glucose Value Tests <70 mg/dL
Time Frame: Up to 10 days
Population: Participants who completed the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of tests
Arm/Group | Adult Cohort - Medtronic Android Interface | Adult Cohort - Integrated System Interface | Adolescent Cohort
Number analyzed (Participants) | 8 | 9 | 14
percentage of tests
  Open loop | 4.7 (5.1) | 13.0 (9.7) | 11.7 (9.9)
  Closed loop | 1.4 (1.7) | 7.6 (2.9) | 13.5 (13.9)

7. Secondary Outcome: Percentage of Time With Sensor Glucose Values <70 mg/DL, Adult Cohorts
Time Frame: Up to 10 days
Population: Data are presented for adult cohorts only.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Adult Cohort - Medtronic Android Interface | Adult Cohort - Integrated System Interface
Number analyzed (Participants) | 8 | 9
percentage of time
  Day (open loop) | 2.7 (1.3) | 7.6 (5.4)
  Day (closed loop) | 1.4 (1.8) | 2.0 (1.4)
  Night (open loop) | 3.5 (4.3) | 8.2 (8.7)
  Night (closed loop) | 1.9 (3.4) | 1.2 (1.7)

8. Secondary Outcome: Percentage of Time With Sensor Glucose Values <70 mg/DL, Adolescent Cohort
Time Frame: Up to 10 days
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Adolescent Cohort
Number analyzed (Participants) | 14
percentage of time
  Day (open loop) | 2.7 [0.8 to 9.2]
  Day (closed loop) | 2.5 [1.7 to 3.5]
  Night (open loop) | 2.5 [0.5 to 4.7]
  Night (closed loop) | 0.7 [0.0 to 4.2]

9. Secondary Outcome: Percentage of Fingerstick Meter Glucose Value Tests >300 mg/dL, Adult Cohort - Medtronic Android Interface
Time Frame: Up to 10 days
Population: Data are presented for the Adult Cohort - Medtronic Android Interface only
Measure: Median (Inter-Quartile Range); unit: percentage of readings
Arm/Group | Adult Cohort - Medtronic Android Interface
Number analyzed (Participants) | 8
percentage of readings
  Open loop | 0.0 [0.0 to 3.3]
  Closed loop | 0.7 [0.0 to 3.6]

10. Secondary Outcome: Percentage of Fingerstick Meter Glucose Value Tests >300 mg/dL, Adult Cohort - Integrated System Interface and Adolescent Cohort
Time Frame: Up to 10 days
Population: Data are presented for the Adult Cohort - Integrated System Interface and the Adolescent Cohort only. Participants who completed the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of readings
Arm/Group | Adult Cohort - Integrated System Interface | Adolescent Cohort
Number analyzed (Participants) | 9 | 14
percentage of readings
  Open loop | 3.0 (4.3) | 8.9 (9.8)
  Closed loop | 3.1 (2.5) | 6.7 (9.2)

ADVERSE EVENTS:
Time Frame: Up to 10 days
Arm/Group | Adult Cohort | Adolescent Cohort
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/15
Other Adverse Events (participants affected / at risk) | 0/9 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Cohort (N=9) | Adolescent Cohort (N=15)
Hypoglycaemia (Endocrine disorders) | 0 (0) | 1 (2) — Hypoglycaemia defined as blood glucose <50 mg/dL

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other